CLINICAL TRIAL: NCT04711811
Title: Individual Patient Expanded Access IND Using HB-adMSCs for the Treatment of Chronic Musculoskeletal Pain.
Brief Title: Individual Patient Expanded Access IND of HB-adMSCs for Chronic Musculoskeletal Pain.
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBCMP01
Record Dates: First submitted 2020-12-28; First posted 2021-01-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; trauma; Pain; Stem Cells; Mesenchymal Stem Cells; Autologous MSCs; MSCs
MeSH Terms: conditions — Chronic Pain; Wounds and Injuries; Pain

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: HB-adMSC — Hope Biosciences adipose derived autologous mesenchymal stem cell product

SUMMARY:
This is an Individual Patient Expanded Access IND providing multiple administrations of HBadMSCs for the treatment of Chronic Musculoskeletal Pain. The study duration is approximately 32 weeks, during that time the study subject will complete 1 screening visit, 6 infusion visits, one follow-up visit without infusion and one end of study visit. Next day telephone follow-up visits will occur following each infusion. Efficacy and safety labs as well as quality of life and VAS scores will be obtained.

DETAILED DESCRIPTION:
Visit 1 - Screening During the screening visit, the principal investigator and/or delegated staff must provide a copy of the IRB-approved informed consent form * to the subject before performing any study procedure.

* IRB must provide a certificate action as proof of approval of the informed consent form.

The study subject should take enough time to read this essential document. If the study subject agrees to participate in the clinical trial, after reading the document, he/she must sign it. By giving his/her signature, study subject allows the principal investigator and/or designated staff to perform the following study procedures:

1. Collection of Medical History.
2. Collection of prior (up to a week before screening) and current medications.
3. Evaluation of Inclusion and Exclusion Criteria.
4. Measurement of Weight in lb. and Height in cm.
5. Collection of vital signs, including respiratory rate, pulse rate SPO2, blood pressure and body temperature.
6. Collection of laboratory samples, including Comprehensive Metabolic Panel, Complete Blood Count and Coagulation Panel, C - reactive protein and Erythrocyte sedimentation rate.
7. Physical Examination by the principal investigator.
8. Video documentation of the subject walking and expressing the level of pain he/she presents at that visit.

Visits 2, 3, 4, 6 and 7. (Infusions 1, 2, 3, 5 and 6) Throughout these visits, the principal investigator and/or delegated staff will perform the following assessments:

1. Update Medical History Form if necessary.
2. Update Concomitant medications list if applicable.
3. Measurement of Weight in lb.
4. Collection of vital signs, including respiratory rate, pulse rate SPO2, blood pressure and body temperature.
5. Completion of study questionaries by the subject.
6. Physical Examination by the principal investigator.
7. Investigational Product Administration:

   * Drug Name: HB-adMSCs
   * Route: Intravenous
   * Dose: 200 million
8. Vital signs monitoring 2 hours post drug exposure. (Every 15 minutes for the first hour (0,15, 30, 45 and 60), and every 30 minutes for the second (90 and 120).
9. 24 hours telephone encounter after Investigational Product Administration to assess incidence of adverse events or serious adverse events.
10. Adverse Events monitoring.

Visit 5 (Infusions 4)

1. Update Medical History Form if necessary.
2. Update Concomitant medications list if applicable.
3. Measurement of Weight in lb.
4. Collection of vital signs, including respiratory rate, pulse rate SPO2, blood pressure and body temperature.
5. Collection of laboratory samples, including Comprehensive Metabolic Panel, Complete Blood Count and Coagulation Panel, C - reactive protein and Erythrocyte sedimentation rate.
6. Completion of study questionaries by the subject.
7. Physical Examination by the principal investigator.
8. Investigational Product Administration:

   * Drug Name: HB-adMSCs
   * Route: Intravenous
   * Dose: 200 million
   * Vital signs monitoring 2 hours post drug exposure. (Every 15 minutes for the first hour (0,15, 30, 45 and 60), and every 30 minutes for the second (90 and 120).
9. 24 hours telephone encounter after Investigational Product Administration to assess incidence of adverse events or serious adverse events.
10. Adverse Events monitoring.

Visit 8 - Phone call Follow Up 1

1. Update Medical History Form if necessary.
2. Update Concomitant medications list if applicable.
3. Adverse Events monitoring.

TREATMENT EXTENSION

After the study subject has completed Visit 7 - Infusion 6, the Principal Investigator will analyze the patient's data to determine if the next series of infusions should be provided. The criteria for making this conclusion are as follows:

* The patient must continue to meet inclusion/exclusion criteria for the study.
* The patient must be experiencing pain as evidenced by the VAS for pain.
* The patient must still be having difficulty in daily physical activities as evidenced by SF36 questionnaire.
* The patient must sign a new informed consent for treatment (s) extension.

Before leaving the infusion center, if the subject is authorized to receive the requested treatment extension, the subject must meet the following discharge criteria:

* Able to ambulate
* Respiration non-labored.
* Alert, oriented.
* SpO2 > 94 % on room air.
* SBP 100 to 139 mmHg & DBP 60 to 89 mmHg
* Heart Rate within normal limits (60 to 100 beats per minute)

Visits 9 and 15 (Infusion 7 and 12)

1. Update Medical History Form if necessary.
2. Update Concomitant medications list if applicable.
3. Measurement of Weight in lb.
4. Collection of vital signs, including respiratory rate, pulse rate SPO2, blood pressure and body temperature.
5. Collection of laboratory samples, including Comprehensive Metabolic Panel, Complete Blood Count and Coagulation Panel, C - reactive protein and Erythrocyte sedimentation rate.
6. Completion of study questionaries by the subject.
7. Physical Examination by the principal investigator.
8. Investigational Product Administration:

   * Drug Name: HB-adMSCs
   * Route: Intravenous
   * Dose: 200 million
   * Vital signs monitoring 2 hours post drug exposure. (Every 15 minutes for the first hour (0,15, 30, 45 and 60), and every 30 minutes for the second (90 and 120).
9. 24 hours telephone encounter after Investigational Product Administration to assess incidence of adverse events or serious adverse events.
10. Adverse Events monitoring.

Visits 10, 11, 13, 14, 16 and 17 (Infusions 8, 9, 10, 11, 13 and 14)

1. Update Medical History Form if necessary.
2. Update Concomitant medications list if applicable.
3. Measurement of Weight in lb.
4. Collection of vital signs, including respiratory rate, pulse rate SPO2, blood pressure and body temperature.
5. Completion of study questionaries by the subject.
6. Physical Examination by the principal investigator.
7. Investigational Product Administration:

   * Drug Name: HB-adMSCs
   * Route: Intravenous
   * Dose: 200 million
   * Vital signs monitoring 2 hours post drug exposure. (Every 15 minutes for the first hour (0,15, 30, 45 and 60), and every 30 minutes for the second (90 and 120).
8. 24 hours telephone encounter after Investigational Product Administration to assess incidence of adverse events or serious adverse events.
9. Adverse Events monitoring.

Visit 12 - Follow Up Visit.

1. Update Medical History Form if necessary.
2. Update Concomitant medications list if applicable.
3. Measurement of Weight in lb.
4. Collection of vital signs, including respiratory rate, pulse rate SPO2, blood pressure and body temperature.
5. Collection of laboratory samples, including Comprehensive Metabolic Panel, Complete Blood Count and Coagulation Panel, C - reactive protein and Erythrocyte sedimentation rate.
6. Completion of study questionaries by the subject.
7. Physical Examination by the principal investigator.
8. Adverse Events monitoring.

Visit 18. (End of Study)

1. Update Medical History Form if necessary.
2. Update Concomitant medications list if applicable.
3. Measurement of Weight in lb.
4. Collection of vital signs, including respiratory rate, pulse rate SPO2, blood pressure and body temperature.
5. Collection of laboratory samples, including Comprehensive Metabolic Panel, Complete Blood Count and Coagulation Panel, C - reactive protein and Erythrocyte sedimentation rate.
6. Completion of study questionaries by the subject.
7. Physical Examination by the principal investigator.
8. Adverse Events monitoring.

ELIGIBILITY:
IND # 27057

Inclusion Criteria:

1. Subject is > 18 years of age at the time of signing the informed consent form.
2. Subject has the diagnosis of chronic musculoskeletal pain for a least 1 year or VAS score > 7 a screening visit.
3. Subject has provided informed consent before initiation of any study procedure.
4. Subject and sexual partner if woman of childbearing potential must use a least 1 highly effective form of birth control* throughout the study and for 6 months after the last dose of the investigational product.

Exclusion Criteria:

1. Subject has any active infection for which antibiotics were indicated within 4 weeks before screening.
2. Subject has known alcoholic addiction or dependency, uses alcohol daily, or has current substance use or abuse.
3. Subject has any active malignancy, including evidence of cutaneous basal, squamous cell carcinoma, or melanoma.
4. Subject has 1 or more significant concurrent medical conditions per investigator judgment, including the following:

   * poorly controlled diabetes.
   * chronic kidney disease
   * heart failure
   * myocardial infarction or unstable angina within 6 months prior to screening.
   * uncontrolled hypertension
5. Subject has received any stem cell treatment within 12 months before first dose of investigational product.
6. Subject has laboratory abnormalities during screening, including the following:

   * White blood cell count < 3000/mm3
   * Platelet count < 125,000mm3
   * Absolute neutrophil count < 1500/mm3
   * Subject has any other laboratory abnormality, which, in the opinion of the investigator poses a safety risk or will prevent the subject for completing the study.
7. Subject is currently receiving treatment in another investigational drug study.
8. Subject is unlikely to complete the study or adhere to the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Djamchid Lotfi, MD, Principal Investigator — Hope Biosciences Stem Cell Research Foundation
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States